CLINICAL TRIAL: NCT01276899
Title: Prospective Study to Identify Molecular Mechanisms of Clinical Resistance to Chemotherapy in Triple Negative Breast Cancer Patients
Brief Title: Study to Identify Molecular Mechanisms of Clinical Resistance to Chemotherapy in Triple Negative Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Jewish General Hospital (Other)
Collaborators: Exactis Innovation (Other); Genome Quebec (Other)
Responsible Party: Principal Investigator, Mark Basik, Principal Investigator, Jewish General Hospital
Other Study IDs: Q-CROC-03
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Triple Negative Breast Cancer
Keywords: Breast Cancer; Triple negative breast cancer; ERnegative, PRnegative and Her2negative; Taxanes; Metastases; Biomarkers; Resistance; Biobanking; Breast cancer with unresectable metastases to the liver; Breast cancer with unresectable metastases to the skin; Breast cancer with unresectable metastases to the lymph node; Neoadjuvant chemotherapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Neoplasm Metastasis | interventions — Biopsy, Large-Core Needle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor samples from the primary breast tumor or metastatic lesions will be obtained by needle core biopsy. In the neoadjuvant setting, samples will be also collected at the time of surgery. To obtain sufficient material for tissue banking, four needle core biopsies will be removed from the same neoplastic lesion. Two of the biospecimens will be snap frozen for phosphoprotein preservation, one will be placed in RNAlater for nucleic acid preservation and the other one will be placed in formalin for FFPE. Additionally, blood samples will be collected at different time points during treatment.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Neoadjuvant setting
  Interventions: Procedure: Needle core biopsies
- Metastatic setting
  Interventions: Procedure: Needle core biopsies of metastatic lesion

INTERVENTIONS:
Procedure: Needle core biopsies — No investigational products will be administered to subjects as part of this translational research study. Needle core biopsies will be done to collect tumor samples.
  A taxane-based regimen will be administered as per the standard of care at each treating institution. Tissue samples from primary tumors will be collected and banked before the start of chemotherapy, after chemotherapy and at the time of surgery. Additionally, blood samples will be drawn before treatment initiation (baseline) and at different time points during treatment and stored in the tissue biobank.
  Groups: Neoadjuvant setting
Procedure: Needle core biopsies of metastatic lesion — No investigational products will be administered to subjects as part of this translational research study. Needle core biopsies will be done to collect metastasis tumor samples.
  Chemotherapy will be administered as per the standard of care at each treating institution. Tissue samples from metastatic tumors lesions will be collected and banked before the start of chemotherapy and at the time of progression. Additionally, blood samples will be drawn before treatment initiation (baseline) and at different time points during treatment and stored in the tissue biobank.
  Groups: Metastatic setting

SUMMARY:
This is a multicenter translational study to understand therapeutic resistance in patients undergoing standard chemotherapy for triple negative breast cancer.

In the neoadjuvant setting, biopsy tissue samples from primary tumor will be collected and banked before the start of chemotherapy and after the completion of the treatment (post-chemotherapy and at the time of surgery). In the metastatic setting, tissue samples from metastatic lesions will be collected and banked before the start of chemotherapy and at the time of tumor progression. Additionally, blood samples will be drawn before treatment initiation (baseline) and at different time points during treatment. All samples will be stored in the Biological Resource Repository.

DETAILED DESCRIPTION:
Mechanisms of resistance have been studied for many years in various experimental models. However, many drugs that are highly effective in experimental models at overcoming resistance have been either ineffective or marginally active in preliminary clinical studies. Thus after decades of study, most reviews of anti-cancer drug resistance still focus largely on experimental models, which may not reflect resistance in humans. However, recent studies have demonstrated that clinical resistance occurs in primary and metastatic tumors that may have undergone significant molecular evolution due to treatment effects and the selection of clones as recently shown in breast cancer.

Triple negative breast cancer is a subtype that carries a poor prognosis and a high incidence of early metastatic recurrence. Furthermore, no target therapy is efficacious up to now in this subtype. Thus, identification of mechanisms of resistance to available therapies and prediction of tumoral response to various treatments could help in the management of patients affected by this particularly aggressive type of breast cancer.

The goals of this study are two-fold. First, to build a biobank of blood and tissue specimens, prior to starting chemotherapy and at a determined time-point (surgery or progression of disease), from patients undergoing the chemotherapeutic treatments in the neoadjuvant and metastatic settings. Second, to use cutting-edge molecular techniques available in several Quebec research centers, to carefully compare these pre and post treatment samples to identify "molecular factors of resistance". The discovery of these factors will help oncologists in triaging patients to receive the most beneficial therapy by recognizing when not to give particular treatment and will be essential for reducing the potential for harmful side effects and for avoiding the extremely high cost of modern treatments when they can be predicted to be ineffective.

ELIGIBILITY:
Inclusion Criteria:

Neoadjuvant setting

1. Histologically confirmed diagnosis of adenocarcinoma of the breast
2. Patient candidate for neoadjuvant chemotherapy (taxane-based)
3. Triple negative (ERnegative, PRnegative and Her2negative as defined by local standards)
4. Normal coagulation profile; including INR/ PTT ≤ 1.5 x ULN.
5. ECOG 0,1 or 2
6. Provide written consent after the investigational nature, study design, risks and benefits of the study have been explained.
7. Able to adhere to the study visit schedule and other protocol requirements.

Metastatic setting

1. Patients with histologically confirmed primary adenocarcinoma of the breast
2. Metastatic (stage IV) disease at initial diagnosis or following previous diagnosis of primary breast cancer
3. At least one metastatic site accessible for biopsy.
4. ER-negative, PgR negative and HER2 negative as per local standards
5. Scheduled to receive chemotherapy for triple negative metastatic breast cancer.
6. Measurable disease (at least one unidimensionally measurable lesion)
7. Normal coagulation profile; including INR/ PTT ≤ 1.5 x ULN.
8. ECOG 0,1 or 2
9. Life expectancy of 12 or more weeks.
10. Provide written consent after the investigational nature, study design, risks and benefits of the study have been explained.
11. Able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

Neoadjuvant setting

1. Positive for ER, PR or Her2 as defined by local standards
2. Clinical or radiological evidence of metastatic disease
3. Inadequate or unusable tissue as the only tissue available for biopsy
4. Other non-malignant systemic disease to preclude treatment with chemotherapy regimen or prevent follow-up
5. Diagnosis of inflammatory breast cancer
6. Known infection with HIV or hepatitis

Metastatic setting

1. Patients with ER+, PR+ or HER2+ tumors demonstrated by local standards
2. Inadequate or unusable tissue as the only tissue available for biopsy
3. Other non-malignant systemic disease to preclude treatment with standard chemotherapy regimen or prevent follow-up
4. Abnormal coagulation profile
5. The planned concurrent administration of therapies (e.g. palliative radiotherapy) that target metastatic sites accessible for biopsy
6. Known infection with HIV or hepatitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in patients with a diagnosis of breast cancer and pathologically identified as triple negative (not expressing estrogen receptor (ER), progesterone receptor (PR) and HER2 protein, and not showing ERBB2 gene amplification) who will be undergoing neoadjuvant treatment or chemotherapy for metastatic disease.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-09 (Actual); Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Biomarkers changes in patients that have been exposed to chemotherapy | 3 years

SECONDARY OUTCOMES:
Create a unique bank of biospecimens from patients with triple negative breast tumors comprising tumor material and plasma collected in a specific and well defined clinical context. | 2 years
Study mechanisms of resistance to chemotherapy by profiling for the first time resistant tumors in both the metastatic and advanced primary tumor settings. | 3 years
Identify biomarkers that will be used as predictors of therapeutic resistance in the tissue and blood of patients with triple negative breast tumors | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Basik, MD, Principal Investigator — Segal Cancer Centre, Jewish General Hospital
Locations (8):
- John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois, United States
- Canada (7):
  - Centre Hospitalier de l'Université de Montréal -- Hotel-Dieu, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal- Notre-Dame, Montreal, Quebec
  - Hôpital Royal Victoria, Montreal, Quebec
  - Hôpital Sacré-Coeur, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - St-Mary's Hospital Center, Montreal, Quebec
  - Hopital du St-Sacrement, Québec